CLINICAL TRIAL: NCT03034824
Title: Comparison Of Er,Cr:YSGG and Diode Laser on the Periodontal Parameters and Cytokines Levels in Patients With Generalized Aggressive Periodontitis
Brief Title: Effects of Er,Cr:YSGG, Diode Lasers on GCF Cytokines Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ahmet Cemil Talmac, PhD, Dr. Dt., Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: JOP-16-0797
Record Dates: First submitted 2016-12-21; First posted 2017-01-27 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Aggressive Periodontitis
Keywords: diode laser; Er,Cr:YSGG laser; Aggressive Periodontitis; Clinical periodontal parameters; Gingival crevicular fluid cytokines levels
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Scaling and root planing (SRP)-Control (Experimental): Only non-surgical initial periodontal treatment (scaling and root planing)
  Interventions: Procedure: Scaling and root planing (SRP)-Control
- SRP+940±15 nm diode laser (Experimental): In addition to non-surgical initial periodontal treatment (scaling and root planing), individuals received 940±15 nm Diode laser
  Interventions: Procedure: SRP+940±15 nm diode laser
- SRP+Er,Cr:YSGG laser (Experimental): In addition to non-surgical initial periodontal treatment (scaling and root planing), individuals received Er,Cr:YSGG laser
  Interventions: Procedure: SRP+Er,Cr:YSGG laser

INTERVENTIONS:
Procedure: SRP+940±15 nm diode laser — In addition to Non-surgical periodontal treatment, the individuals diagnosed with Generalized Aggressive Periodontitis were applied the 940±15 nm diode laser.
  Arms: SRP+940±15 nm diode laser
Procedure: SRP+Er,Cr:YSGG laser — In addition to Non-surgical periodontal treatment, the individuals diagnosed with Generalized Aggressive Periodontitis were applied the Er,Cr:YSGG laser.
  Arms: SRP+Er,Cr:YSGG laser
Procedure: Scaling and root planing (SRP)-Control — Only Non-surgical periodontal treatment
  Arms: Scaling and root planing (SRP)-Control

SUMMARY:
The aim of our study is to determine the interleukin-1βeta (IL-1β), interleukin-8 (IL-8) and tumor necrosis factor-αlfa (Tnf-α) levels in gingival crevicular fluid (GCF) and clinical periodontal parameters following the treatment with Erbium,Chromium:Yttrium-Scandium-Gallium-Garnet (Er,Cr:YSGG) and diode lasers in adjunct to scaling and root planing (SRP) in patients with generalized aggressive periodontitis (GAgP). Twenty-six patients with GAgP (n=26) were enrolled in the study. The study was designed as a "split-mouth" study. In each patient, three quadrants were randomly determined as SRP-control, SRP+Er,Cr:YSGG and SRP+Diode laser. Clinical periodontal measurements were recorded at the baseline and third month after the treatment. Cytokines levels in GCF were determined by enzyme-linked immunosorbent assay (ELISA).

DETAILED DESCRIPTION:
A total of 26 individuals were included in our study. Diagnoses were made after the clinical and radiographic examinations on patients who applied to the Yuzuncu Yil University Faculty of Dentistry, Department of Periodontology Clinics in 2014-2015. It was ensured that the individuals who were included in the study did not have any systemic diseases; were not menopausal, pregnant or lactating; had not used antibiotics or any other medication affecting the immune system in the previous six months; were non-smokers; had at least 16 teeth in their mouth; and had not received any periodontal treatment in the previous 6 months. The subjects involved in the study were told the aim and content of the study by a clinician, and they signed an approval form stating that they voluntarily participated in the survey. Each individual read the Helsinki Declaration before joining the study. The Human Ethics Research Committee of Yuzuncu Yil University (no.B.30.2.YYU.0.01.00.00/44-100912) gave the approval to carry out the study.

The including criteria were applied in diagnosing generalized aggressive periodontitis (International Workshop for Classification of Periodontal Diseases in 1999). Clinical periodontal assessments, including periodontal status, were conducted by measuring the bleeding on probing (BOP), plaque index (PI), gingival index (GI), probing pocket depth (PPD) and clinical attachment level (CAL) at 6 sites per tooth by another clinician. The clinical periodontal indices measured during the research were evaluated site-specifically by including the mesial and distal of those teeth from which GCF samples were obtained.

All individuals received non-surgical initial periodontal treatment. At the baseline of the study all quadrants were shown the similarity of periodontal disease. The procedures outlined below were applied to all individuals in the study in randomly selected three different quadrants. The study was designed as a "split-mouth" study.

1. Only SRP group (SRP-Control)
2. SRP+Er,Cr:YSGG laser group (SRP+Er,Cr:YSGG)
3. SRP+940±15 nm diode laser group (SRP+Diode) GCF sample sites were selected after probing measurements were taken. The GCF samples were collected at the baseline of the study and on the 3rd month following treatment. The GCF samples were taken from the deepest pocket in all quadrants. The samples were collected with paper strips (Periopaper Oraflow, NewYork, USA) that were cut in standard size. Before the sampling procedure, supragingival plaque was removed and then the sites were isolated from saliva with sterile buffer and sterile cotton rolls. The sampled tooth surfaces were dried by slightly blowing air on them. The paper strips were inserted until a light resistance in the sulcus was felt, and they were left there for 30 seconds. The strips that were contaminated with blood were not included in the evaluation. The fluid amount was measured by a Periotron device (Periotron 8000, Oraflow, NewYork, USA) and was converted to GCF volume in ml units. The four strips which were obtained from every patient were placed into individual Eppendorf tubes, each of which contained 500 μl of liquid (Phosphate Buffer Saline (PBS)-pH 7.4) and a paper strip and were stored at -80o C.

SRP was first performed to the control quadrants of the individuals diagnosed with GAgP; following the SRP procedure, the Er,Cr:YSGG laser was applied. The 940±15 nm diode laser was applied prior to SRP, unlike the Er,Cr:YSGG laser (to prevent changing the diode laser efficiency following bleeding). In the study, the Er,Cr:YSGG laser (Waterlase, Biolase, Irvine, CA, USA) and the 940±15 nm diode laser (Ilase, Biolase, Irvine, CA, USA) were used. For the Er,Cr:YSGG laser, a 14-mm Z-6 tip (600 μm fiberoptic tip, suitable for periodontal use) marked to the depth of the pocket was used at a setting of 10 Hz, 1.5 W (150 mJ), 65% air, 55% water with H mode, 140 μs pulse length. The total irradiation time was 30 s. The 940±15 nm diode laser with MZ6-14 mm standard tip was used at a setting in continuous wave mode. The irradiation times for 940±15 nm diode laser were adjusted to 20 s.

The TNF-α, IL-1β and IL-8 analysis in GCF was conducted through the ELISA method by means of commercial ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* No systemic diseases
* Not used antibiotics or any other medication affecting the immune system in the previous six months
* Non-smokers
* Have at least 16 teeth in their mouth
* Have not received any periodontal treatment in the previous 6 months

Exclusion Criteria:

* Under 18 age
* Pregnant women

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Periodontal Clinical Indices | 1 year
  Bleeding on probing
Periodontal Clinical Indices | 1 year
  Plaque index
Periodontal Clinical Indices | 1 year
  Gingival index
Periodontal Clinical Indices | 1 year
  Probing pocket depth
Periodontal Clinical Indices | 1 year
  Clinical attachment level

SECONDARY OUTCOMES:
Cytokines levels in gingival crevicular fluids | 1 year
  Interleukin-1β
Cytokines levels in gingival crevicular fluids | 1 year
  Interleukin-8
Cytokines levels in gingival crevicular fluids | 1 year
  Tumor necrosis factor-α

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet C Talmac, PhD, Principal Investigator — Researcher

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hakki SS, Korkusuz P, Berk G, Dundar N, Saglam M, Bozkurt B, Purali N. Comparison of Er,Cr:YSGG laser and hand instrumentation on the attachment of periodontal ligament fibroblasts to periodontally diseased root surfaces: an in vitro study. J Periodontol. 2010 Aug;81(8):1216-25. doi: 10.1902/jop.2010.090715. PMID 20476883